CLINICAL TRIAL: NCT02262728
Title: A Phase 2 Open-label Study to Investigate the Efficacy, Safety and Pharmacokinetics of 12 Weeks of Treatment With Simeprevir, Daclatasvir and Sofosbuvir, Followed by a 5-Year Post-treatment Long-term Follow-up, in Treatment-naïve and Treatment-experienced Subjects With Chronic Hepatitis C Virus Genotype 1 or 4 Infection and Decompensated Liver Disease
Brief Title: An Efficacy, Safety and Pharmacokinetics Study of Simeprevir, Daclatasvir and Sofosbuvir in Participants With Chronic Hepatitis C Virus Genotype 1 or 4 Infection and Decompensated Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR105028; TMC435HPC2010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Simeprevir; Daclatasvir; Sofosbuvir; Decompensated Liver Disease
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Panel 1 (Experimental): Participants with Child-Pugh score <7 with evidence of portal hypertension (confirmed by presence of esophageal varices or hepatic venous pressure gradient [HVPG] greater than or equal to 10 millimeter of mercury [mm Hg]) will receive simeprevir (150 milligram [mg] capsule), daclatasvir (60 mg tablet) and sofosbuvir (400 mg tablet) orally once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Daclatasvir; Drug: Sofosbuvir
- Panel 2 (Experimental): Participants with Child-Pugh score 7 to 9 (extremes included) will receive simeprevir (150 mg capsule), daclatasvir (60 mg tablet) and sofosbuvir (400 mg tablet) orally once daily for 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Daclatasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — Simeprevir 150 milligram (mg) capsule orally once daily for 12 weeks
  Other Names: TMC435
Drug: Daclatasvir — Daclatasvir 60 mg tablet orally once daily for 12 weeks
  Other Names: BMS-790052
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet orally once daily for 12 weeks
  Other Names: GS-7977

SUMMARY:
The purpose of this study is to assess the efficacy of a 12-week regimen containing simeprevir, daclatasvir and sofosbuvir in participants with decompensated liver disease (the liver function is insufficient) due to genotype 1 or 4 Hepatitis (inflammation of the liver) C virus (HCV) infection by assessing sustained virologic response 12-weeks after the end of study drug treatment (SVR12).

DETAILED DESCRIPTION:
This is an open-label (all people know which treatment the participants receive) Phase 2 study to investigate the efficacy, safety and pharmacokinetics of simeprevir, daclatasvir and sofosbuvir in treatment-naive (participants have never received HCV treatment with any approved or investigational agent) and treatment - experienced (participants have failed at least one previous course of [Pegylated] interferon [(Peg)IFN], with or without Ribavirin) participants. Participants will be assigned to 1 of 2 panels: Panel 1 (n=20): Child-Pugh score less than (<) 7 with evidence of portal hypertension (confirmed by presence of esophageal varices or HVPG greater than or equal to [>=] 10 mm Hg); Panel 2 (n=20): Child-Pugh score 7 to 9 (extremes included). The total study duration for each participant will be approximately 276 weeks. The study will consist of 3 parts: Screening Phase (approximately 4 weeks) and open-label treatment Phase (from Week 4 to 16) and follow-up Phase (until 5 years after the actual end of study drug treatment). Participants will receive simeprevir (150 milligram [mg] capsule), daclatasvir (60 mg tablet) and sofosbuvir (400 mg tablet) orally once daily for 12 weeks. Efficacy will be primarily evaluated by percentage of participants with SVR12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic Hepatitis C virus (HCV) infection: diagnosis of HCV more than (>) 6 months before the Screening visit, either by detectable HCV ribonucleic acid (RNA), a HCV positive antibody or the presence of histological changes consistent with chronic hepatitis
* HCV genotype 1 or 4 infection and HCV RNA plasma level >10,000 international unit per milliliter (IU/mL) (both determined at screening)
* Presence of cirrhosis, which is defined as a FibroScan with a result of >14.5 kilopascals (kPa) at Screening
* HCV treatment-naive participants: participant has not received treatment with any approved or investigational drug for the treatment of HCV infection and HCV treatment-experienced participants: participant has had at least 1 documented previous course of a non-direct-acting antiviral agent (DAA), interferon (IFN)-based HCV therapy (with or without Ribavirin [RBV]). Last dose in this previous course should have occurred at least 2 months prior to Screening
* Decompensated liver disease: Panel 1: Child Pugh A (mild hepatic impairment) with evidence of portal hypertension [confirmed by the presence of esophageal varices on gastroscopy or hepatic venous pressure gradient (HVPG) greater than or equal to (>=) 10 millimeter of mercury (mm Hg)], Panel 2: Child-Pugh B (moderate hepatic impairment) 7 to 9 (extremes included)

Exclusion Criteria:

* Co-infection with any HCV genotype
* Co-infection with human immunodeficiency virus (HIV)-1 or -2 (positive HIV-1 or HIV-2 antibodies test at Screening)
* Co-infection with hepatitis B virus (hepatitis B surface antigen [HBsAg] positive)
* Any evidence of liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A infection, drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HCV liver disease considered clinically significant by the Investigator
* Use of any disallowed therapies before the planned first dose of study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- San Antonio, Texas, United States

REFERENCES:
- [Derived] Lawitz E, Poordad F, Gutierrez JA, Beumont M, Beets G, Vandevoorde A, Remoortere PV, Luo D, Vijgen L, Eygen VV, Gamil M. Simeprevir, daclatasvir, and sofosbuvir for hepatitis C virus-infected patients: Long-term follow-up results from the open-label, Phase II IMPACT study. Health Sci Rep. 2020 Feb 22;3(2):e145. doi: 10.1002/hsr2.145. eCollection 2020 Jun. PMID 32270053
- [Derived] Lawitz E, Poordad F, Gutierrez JA, Kakuda TN, Picchio G, Beets G, Vandevoorde A, Van Remoortere P, Jacquemyn B, Luo D, Ouwerkerk-Mahadevan S, Vijgen L, Van Eygen V, Beumont M. Simeprevir, daclatasvir and sofosbuvir for hepatitis C virus-infected patients with decompensated liver disease. J Viral Hepat. 2017 Apr;24(4):287-294. doi: 10.1111/jvh.12645. Epub 2016 Nov 23. PMID 27878906

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel 1 SMV 150mg/DCV 60mg/SOF 400mg: Participants with Child-Pugh score <7 with evidence of portal hypertension (confirmed by presence of esophageal varices or hepatic venous pressure gradient [HVPG] greater than or equal to 10 millimeters of mercury [mm Hg]) received simeprevir (150 milligram [mg] capsule), daclatasvir (60 mg tablet) and sofosbuvir (400 mg tablet) orally once daily for 12 weeks.
- Panel 2 SMV 150mg/DCV 60mg/SOF 400mg: Participants with Child-Pugh score 7 to 9 (extremes included) received simeprevir (150 mg capsule), daclatasvir (60 mg tablet) and sofosbuvir (400 mg tablet) orally once daily for 12 weeks.
Period: Treatment Period (12 Weeks)
Arm/Group | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg
Started | 19 | 21
Completed | 19 (Participants who completed continued follow-up phase.) | 21 (Participants who completed continued follow-up phase.)
Not Completed | 0 | 0
Period: Follow-up Phase (3 Years)
Arm/Group | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg
Started | 19 | 21
Completed | 15 | 18
Not Completed | 4 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 64] | 61 [50 to 75] | 58.5 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 14 | 11 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After End of Study Drug Treatment (SVR12)
Description: Participants were considered to have achieved SVR12 if the hepatitis C virus ribonucleic acid (HCV RNA) was less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detectable or undetectable at 12 weeks after the end of study drug treatment.
Time Frame: Week 24
Population: The intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A: Participants with Child-Pugh score <7 with evidence of portal hypertension (confirmed by presence of esophageal varices or hepatic venous pressure gradient [HVPG] greater than or equal to 10 millimeter of mercury [mm Hg]) received simeprevir (SMV) (150 milligram [mg] capsule), daclatasvir (DCV) (60 mg tablet) and sofosbuvir (SOF) (400 mg tablet) orally once daily for 12 weeks.
- SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B: Participants with Child-Pugh score 7 to 9 (extremes included) received simeprevir (SMV) (150 mg capsule), daclatasvir (DCV) (60 mg tablet) and sofosbuvir (SOF) (400 mg tablet) orally once daily for 12 weeks.
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Percentage of Participants | 100 [82.4 to 100] | 100 [83.9 to 100]

2. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Response
Description: On-treatment virologic response was determined by HCV RNA results satisfying a specified threshold. The following thresholds were considered at any time point: <LLOQ undetectable, <LLOQ detectable, and <LLOQ undetectable or detectable. The LLOQ value was 15 IU/mL. Very rapid virologic response (vRVR) is undetectable HCV RNA at Week 2 while on treatment and Rapid virologic response (RVR) is undetectable HCV RNA at Week 4 while on treatment.
Time Frame: Week 1, 2, 4, 6, 8, 10, 12
Population: The intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug. Here, 'n' signifies number of participants evaluable for this outcome measure at specific time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Percentage of Participants
  Week 1 : >= 15 IU/mL: number analyzed (Participants) | 18 | 21
  Week 1 : >= 15 IU/mL | 72.2 | 76.2
  Week 1 : < 100 IU/mL: number analyzed (Participants) | 18 | 21
  Week 1 : < 100 IU/mL | 61.1 | 38.1
  Week 1: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 18 | 21
  Week 1: < 15 IU/mL undetect/detectable | 27.8 | 23.8
  Week 1 : < 15 IU/mL detectable: number analyzed (Participants) | 18 | 21
  Week 1 : < 15 IU/mL detectable | 11.1 | 19.0
  Week 1 : < 15 IU/mL Undetectable: number analyzed (Participants) | 18 | 21
  Week 1 : < 15 IU/mL Undetectable | 16.7 | 4.8
  Week 2 : >= 15 IU/mL | 10.5 | 47.6
  Week 2 : < 100 IU/mL | 94.7 | 71.4
  Week 2: < 15 IU/mL undetect/detectable | 89.5 | 52.4
  Week 2 : < 15 IU/mL detectable | 36.8 | 19.0
  Week 2: < 15 IU/mL undetectable (vRVR) | 52.6 | 33.3
  Week 4 : >= 15 IU/mL: number analyzed (Participants) | 18 | 21
  Week 4 : >= 15 IU/mL | 0 | 9.5
  Week 4 : < 100 IU/mL: number analyzed (Participants) | 18 | 21
  Week 4 : < 100 IU/mL | 100.0 | 100.0
  Week 4: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 18 | 21
  Week 4: < 15 IU/mL undetect/detectable | 100.0 | 90.5
  Week 4 : < 15 IU/mL detectable: number analyzed (Participants) | 18 | 21
  Week 4 : < 15 IU/mL detectable | 5.6 | 28.6
  Week 4 : < 15 IU/mL undetectable (RVR): number analyzed (Participants) | 18 | 21
  Week 4 : < 15 IU/mL undetectable (RVR) | 94.4 | 61.9
  Week 6 : >= 15 IU/mL: number analyzed (Participants) | 19 | 20
  Week 6 : >= 15 IU/mL | 0 | 0
  Week 6 : < 100 IU/mL: number analyzed (Participants) | 19 | 20
  Week 6 : < 100 IU/mL | 100.0 | 100.0
  Week 6: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 19 | 20
  Week 6: < 15 IU/mL undetect/detectable | 100.0 | 100.0
  Week 6 : < 15 IU/mL detectable: number analyzed (Participants) | 19 | 20
  Week 6 : < 15 IU/mL detectable | 5.3 | 20.0
  Week 6 : < 15 IU/mL undetectable: number analyzed (Participants) | 19 | 20
  Week 6 : < 15 IU/mL undetectable | 94.7 | 80.0
  Week 8 : >= 15 IU/mL: number analyzed (Participants) | 18 | 21
  Week 8 : >= 15 IU/mL | 0 | 0
  Week 8 : < 100 IU/mL: number analyzed (Participants) | 18 | 21
  Week 8 : < 100 IU/mL | 100.0 | 100.0
  Week 8: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 18 | 21
  Week 8: < 15 IU/mL undetect/detectable | 100.0 | 100.0
  Week 8 : < 15 IU/mL detectable: number analyzed (Participants) | 18 | 21
  Week 8 : < 15 IU/mL detectable | 0 | 4.8
  Week 8 : < 15 IU/mL undetectable: number analyzed (Participants) | 18 | 21
  Week 8 : < 15 IU/mL undetectable | 100.0 | 95.2
  Week 10 : >= 15 IU/mL: number analyzed (Participants) | 18 | 21
  Week 10 : >= 15 IU/mL | 0 | 0
  Week 10 : < 100 IU/mL: number analyzed (Participants) | 18 | 21
  Week 10 : < 100 IU/mL | 100.0 | 100.0
  Week 10: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 18 | 21
  Week 10: < 15 IU/mL undetect/detectable | 100.0 | 100.0
  Week 10 : < 15 IU/mL detectable: number analyzed (Participants) | 18 | 21
  Week 10 : < 15 IU/mL detectable | 0 | 0
  Week 10 : < 15 IU/mL undetectable: number analyzed (Participants) | 18 | 21
  Week 10 : < 15 IU/mL undetectable | 100.0 | 100.0
  Week 12 : >= 15 IU/mL: number analyzed (Participants) | 17 | 19
  Week 12 : >= 15 IU/mL | 0 | 0
  Week 12 :< 100 IU/mL: number analyzed (Participants) | 17 | 19
  Week 12 :< 100 IU/mL | 100.0 | 100.0
  Week 12: < 15 IU/mL undetect/detectable: number analyzed (Participants) | 17 | 19
  Week 12: < 15 IU/mL undetect/detectable | 100.0 | 100.0
  Week 12 : < 15 IU/mL detectable: number analyzed (Participants) | 17 | 19
  Week 12 : < 15 IU/mL detectable | 0 | 0
  Week 12 : < 15 IU/mL undetectable: number analyzed (Participants) | 17 | 19
  Week 12 : < 15 IU/mL undetectable | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With SVR 4 Weeks After End of Study Drug Treatment (SVR4) and SVR 24 Weeks After End of Study Drug Treatment (SVR24)
Description: Participants were considered to have achieved SVR4 and SVR24 if the HCV RNA was <LLOQ detectable or undetectable at 4 weeks and 24 weeks respectively after the end of study drug treatment. The LLOQ value was 15 IU/mL.
Time Frame: Week 16 and Week 36
Population: The intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug. Here , 'n' signifies number of participants evaluable for this outcome measure at specific time point.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Percentage of Participants
  SVR 4 | 100 [82.4 to 100] | 100 [83.9 to 100]
  SVR 24: number analyzed (Participants) | 19 | 9
  SVR 24 | 100 [82.4 to 100] | 100 [NA to NA] — 95% Confidence Interval was not calculated since less than 10 participants were evaluable for the specific arm group.

4. Secondary Outcome: Percentage of Participants With HCV NS3/4A Sequence, NS5A and NS5B After End of Treatment in Participants Not Achieving SVR
Description: Sequencing of the HCV nonstructural protein 3/4A (NS3/4A), nonstructural protein 5A (NS5A) and nonstructural protein 5B (NS5B) genes was done to identify pre-existing sequence polymorphisms and characterize emerging HCV viral variants in participants not achieving SVR. All participants in this study achieved SVR12. Therefore, reasons for not achieving SVR12 are not applicable.
Time Frame: Baseline, Day 3, Week 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and Year 1, 1.5, 2, 2.5, 3 after end of treatment
Population: The ITT analysis set who failed achieving SVR. Since all participants achieved SVR, the number of participants for this endpoint analysis was zero.
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Absolute Values of Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) Levels at Follow-up Week 24 (Week 36)
Time Frame: Follow-up Week 24 (Week 36)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Units per Liter (U/L)
  Baseline : ALT | 137.8 (101.90) | 60.9 (29.52)
  Baseline : AST | 119.1 (80.57) | 83.5 (35.68)
  Follow-Up Week 24 : ALT: number analyzed (Participants) | 18 | 9
  Follow-Up Week 24 : ALT | 34.8 (11.30) | 32.3 (9.75)
  Follow-Up Week 24 : AST: number analyzed (Participants) | 18 | 9
  Follow-Up Week 24 : AST | 39.2 (21.86) | 35.0 (10.31)

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Simeprevir, Daclatasvir, Sofosbuvir and GS-331007 (Sofosbuvir Metabolite)
Description: Tmax is the time to reach maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose on Weeks 2 and 8
Population: Pharmacokinetic (PK) analysis set included all participants who received atleast 1 dose of study drug and had valid pharmacokinetic profile. Here 'n' signifies number of participants analyzed for this outcome measure at specific time point.
Measure: Median (Full Range); unit: Hours
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Hours
  Simeprevir: Week 2 | 6.00 [4.00 to 12.00] | 8.00 [2.00 to 24.00]
  Simeprevir: Week 8: number analyzed (Participants) | 18 | 20
  Simeprevir: Week 8 | 6.00 [3.00 to 12.00] | 8.00 [0.50 to 24.00]
  Daclatasvir: Week 2: number analyzed (Participants) | 18 | 21
  Daclatasvir: Week 2 | 3.00 [0.50 to 6.00] | 4.00 [1.00 to 8.00]
  Daclatasvir: Week 8: number analyzed (Participants) | 18 | 21
  Daclatasvir: Week 8 | 2.50 [0.00 to 8.00] | 4.00 [0.00 to 12.00]
  Sofosbuvir: Week 2: number analyzed (Participants) | 18 | 21
  Sofosbuvir: Week 2 | 1.00 [0.50 to 4.00] | 2.00 [0.50 to 4.08]
  Sofosbuvir: Week 8: number analyzed (Participants) | 18 | 21
  Sofosbuvir: Week 8 | 1.75 [0.50 to 12.00] | 2.00 [1.00 to 6.00]
  GS-331007: Week 2: number analyzed (Participants) | 18 | 21
  GS-331007: Week 2 | 4.00 [1.50 to 4.17] | 4.00 [1.50 to 8.00]
  GS-331007: Week 8: number analyzed (Participants) | 18 | 21
  GS-331007: Week 8 | 4.00 [2.00 to 12.00] | 4.00 [3.00 to 8.00]

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours After Dosing (AUC[0-24]) of Simeprevir, Daclatasvir, Sofosbuvir and GS-331007 (Sofosbuvir Metabolite)
Description: The AUC(0-24) is area under the plasma concentration-time curve from time 0 to 24 hours after dosing.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose on Weeks 2 and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
ng.h/mL
  Simeprevir : Week 2 | 113835 (91598) | 142162 (80217)
  Simeprevir : Week 8: number analyzed (Participants) | 18 | 20
  Simeprevir : Week 8 | 98568 (80037) | 207221 (162168)
  Daclatasvir : Week 2: number analyzed (Participants) | 18 | 21
  Daclatasvir : Week 2 | 16487 (6323) | 17858 (7726)
  Daclatasvir : Week 8: number analyzed (Participants) | 18 | 21
  Daclatasvir : Week 8 | 15574 (5347) | 20787 (10741)
  Sofosbuvir : Week 2: number analyzed (Participants) | 18 | 21
  Sofosbuvir : Week 2 | 2870 (978) | 3915 (1258)
  Sofosbuvir : Week 8: number analyzed (Participants) | 18 | 21
  Sofosbuvir : Week 8 | 2746 (963) | 3933 (1315)
  GS-331007 : Week 2: number analyzed (Participants) | 18 | 21
  GS-331007 : Week 2 | 17900 (6320) | 21118 (11301)
  GS-331007 : Week 8: number analyzed (Participants) | 18 | 21
  GS-331007 : Week 8 | 18132 (7469) | 22829 (15394)

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Simeprevir, Daclatasvir, Sofosbuvir and GS-331007 (Sofosbuvir Metabolite)
Description: The Cmax is the maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose on Weeks 2 and 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
nanogram per milliliter (ng/mL)
  Simeprevir : Week 2 (reference) | 6976 (4439) | 7726 (3946)
  Simeprevir : Week 8 (test): number analyzed (Participants) | 18 | 20
  Simeprevir : Week 8 (test) | 6029 (3936) | 10498 (7492)
  Daclatasvir : Week 2: number analyzed (Participants) | 18 | 21
  Daclatasvir : Week 2 | 1187 (397) | 1145 (440)
  Daclatasvir : Week 8: number analyzed (Participants) | 18 | 21
  Daclatasvir : Week 8 | 1072 (313) | 1210 (543)
  Sofosbuvir : Week 2: number analyzed (Participants) | 18 | 21
  Sofosbuvir : Week 2 | 1571 (738) | 1615 (986)
  Sofosbuvir : Week 8: number analyzed (Participants) | 18 | 21
  Sofosbuvir : Week 8 | 1276 (856) | 1527 (993)
  GS-331007 : Week 2: number analyzed (Participants) | 18 | 21
  GS-331007 : Week 2 | 1403 (369) | 1561 (720)
  GS-331007 : Week 8: number analyzed (Participants) | 18 | 21
  GS-331007 : Week 8 | 1404 (361) | 1594 (952)

9. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Simeprevir, Daclatasvir, Sofosbuvir and GS-331007 (Sofosbuvir Metabolite)
Description: The Cmin is the minimum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose on Weeks 2 and 8
Population: PK analysis set included all participants who received atleast 1 dose of study drug and had valid pharmacokinetic profile. Here 'n' signifies number of participants analyzed for this outcome measure at specific time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
ng/mL
  Simeprevir : Week 2 | 3133 (3410) | 4363 (3081)
  Simeprevir : Week 8: number analyzed (Participants) | 18 | 20
  Simeprevir : Week 8 | 2639 (2725) | 6955 (6035)
  Daclatasvir : Week 2 | 414 (230) | 519 (275)
  Daclatasvir : Week 8: number analyzed (Participants) | 18 | 21
  Daclatasvir : Week 8 | 442 (192) | 660 (416)
  Sofosbuvir : Week 2 | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL]) | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL])
  Sofosbuvir : Week 8: number analyzed (Participants) | 18 | 21
  Sofosbuvir : Week 8 | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL]) | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/milliliter[ng/mL])
  GS-331007 : Week 2 | 419 (198) | 441 (254)
  GS-331007 : Week 8: number analyzed (Participants) | 18 | 21
  GS-331007 : Week 8 | 443 (213) | 523 (392)

10. Secondary Outcome: Pre-dose (Trough) Concentration (C0h) of Simeprevir, Daclatasvir, Sofosbuvir and GS-331007 (Sofosbuvir Metabolite)
Description: The C0h is the pre-dose plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours post-dose on Weeks 2 and 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
nanogram/milliliter (ng/mL)
  Simeprevir : Week 2 | 3577 (3685) | 5218 (3461)
  Simeprevir : Week 8: number analyzed (Participants) | 16 | 21
  Simeprevir : Week 8 | 3160 (3725) | 8577 (7398)
  Daclatasvir : Week 2 | 494 (279) | 646 (384)
  Daclatasvir : Week 8: number analyzed (Participants) | 16 | 21
  Daclatasvir : Week 8 | 492 (232) | 824 (476)
  Sofosbuvir : Week 2 | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL]) | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL])
  Sofosbuvir : Week 8: number analyzed (Participants) | 16 | 21
  Sofosbuvir : Week 8 | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL]) | NA (NA) — Data was not reported as participants had concentration below the limit of quantification (less than [<]5.00 nanogram/millilter [ng/mL])
  GS-331007 : Week 2 | 484 (236) | 490 (282)
  GS-331007 : Week 8: number analyzed (Participants) | 16 | 21
  GS-331007 : Week 8 | 478 (262) | 572 (450)

11. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure is defined as participants who do not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of study drug treatment.
Time Frame: Week 12
Population: The intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug. Here "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Percentage of Participants | 0 | 0

12. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse is defined as participants who do not achieve SVR12, with undetectable HCV RNA at the actual end of study drug treatment and confirmed HCV RNA greater than or equal to (>=) LLOQ (15 IU/mL) at Week 16, 24 or 36.
Time Frame: Week 16, 24 and 36
Population: The ITT analysis set who failed achieving SVR. Since all participants achieved SVR, the number of participants for this endpoint (viral relapse) analysis was zero.
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With SVR12 Who Maintained to Have HCV RNA <LLOQ Until the End of 3 Years Follow up
Description: Percentage of participants with SVR12 who maintained to have HCV RNA <LLOQ (15 IU/mL) until the end of 3 years follow up were reported.
Time Frame: Week 24 post treatment until the end of 3-year follow-up
Population: The intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh A | SMV 150mg/DCV 60mg/SOF 400mg - Child-Pugh B
Number analyzed (Participants) | 19 | 21
Percentage of participants | 78.9 | 85.7

ADVERSE EVENTS:
Arm/Group | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg
Serious Adverse Events (participants affected / at risk) | 4/19 | 10/21
Other Adverse Events (participants affected / at risk) | 12/19 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg (N=19) | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg (N=21)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Biliary Dyskinesia (Hepatobiliary disorders) | 0 | 1
Hepatic Lesion (Hepatobiliary disorders) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panel 1 SMV 150mg/DCV 60mg/SOF 400mg (N=19) | Panel 2 SMV 150mg/DCV 60mg/SOF 400mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Irritability (Psychiatric disorders) | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 3
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 4
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Irritability (Psychiatric disorders) | 1 | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Mass (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.